CLINICAL TRIAL: NCT02329197
Title: Intrauterine Injection of Human Chorionic Gonadotropin Before Embryo Transfer in Women With Previous IVF Failure
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Gibreel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H005
Record Dates: First submitted 2014-12-26; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Infertility; Invitro Fertilization
Keywords: Infertility; Invitro fertilization
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): women undergoing IVF treatment will be subjected for intrauterine injection of 10 IU of human chorionic gonadotropin (HCG) (diluted in 0.025ml of tissue culture), 10 minutes before embryo transfer procedure.
  Interventions: Drug: Human Chorionic Gonadotropin (HCG)
- Group B (No Intervention): women undergoing IVF treatment will embryo transfer procedure performed in the standard way without intrauterine injection of HCG.

INTERVENTIONS:
Drug: Human Chorionic Gonadotropin (HCG) — intrauterine injection of HCG prior to embryo transfer in an IVF cycle
  Other Names: u-hCG
  Arms: Group A

SUMMARY:
Women with history of previous IVF cycle failure will be subjected to a fresh IVF cycle. At the time they will be undergoing embryo transfer, 50 IU of human chorionic gonadotropins diluted in 0.025ml of tissue culture media will be injected intrauterine by embryo transfer catheter 10 minutes before embryo transfer procedure.

DETAILED DESCRIPTION:
Infertile women with history of previous IVF cycle failure will be subjected top a fresh IVF cycle. Following controlled ovarian hyperstimulation, ovum pick up and at the time they will be undergoing embryo transfer, 50 IU of human chorionic gonadotropins diluted in 0.025ml of tissue culture media will be injected intrauterine by embryo transfer catheter 10 minutes before embryo transfer procedure.

ELIGIBILITY:
Inclusion Criteria:

- women with previous IVF failure undergoing fresh IVF cycle

Exclusion Criteria:

* women with hydrosalpinges women with intrauterine lesion like submucous fibroid or polyps

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 380 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Live Birth | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Gibreel, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University Teaching Hospital, Al Mansurah, Egypt